CLINICAL TRIAL: NCT02440087
Title: Evaluation of the Dietary Supplement Refill Bypass Administered Sublingually to Reduce Nutritional Deficiencies of Patients Who Underwent Bariatric Surgery Type Gastric Bypass
Brief Title: Evaluation of the Dietary Supplement Refill Bypass to Reduce Nutritional Deficiencies of Patients Who Underwent Bariatric Surgery
Acronym: Refill
Status: Completed | Type: Observational
Sponsor: Refill France (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Other Study IDs: Refill
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Refill Bypass — Dietary supplement

SUMMARY:
This is a cohort, observational, prospective, multicenter, longitudinal study. 100 patients will be followed postoperatively for a period of 12 months. Intermediate statistical analyzes will be performed at 1 month, 3 months, 6 months and 9 months.

This observational study is non-interventional, it does not change the usual care of patients who underwent a bariatric surgery. Data collection will be carried out during routine visits planned in the post-operation usual follow-up. The blood tests are part of the patient's usual care for his bariatric surgery.

Surgeons will include patients for whom they have freely decided to use the dietary supplement Refill under the care of the treatment of obesity. The motivation of the patient and his commitment to the project is evaluated by the surgeon.

The main objective is to evaluate the efficacy of the dietary supplement Refill.

The primary endpoint is the reduction of iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a scheduled bariatric surgery "gastric bypass",
* Patient who performed a blood test before surgery,
* Patient compliant.

Exclusion Criteria:

* Allergy to components of the dietary supplement,
* Pregnancy or breastfeeding,
* Any biological abnormality considered by the investigator significant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients who underwent bariatric surgery
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Reduction of iron deficiency | Month 1, Month 3, Month 6, Month 12 after surgery

SECONDARY OUTCOMES:
Satisfaction questionnaire | Month 1, Month 3, Month 6, Month 12 after surgery
Measurement of Ferritin | Month 3, Month 6, Month 12 after surgery
Measurement of Vitamin B1 | Month 3, Month 6, Month 12 after surgery
Measurement of Vitamin B6 | Month 3, Month 6, Month 12 after surgery
Measurement of Vitamin B9 | Month 3, Month 6, Month 12 after surgery
Measurement of Vitamin B12 | Month 3, Month 6, Month 12 after surgery
Measurement of Hemoglobin | Month 3, Month 6, Month 12 after surgery
Measurement of Albumin | Month 3, Month 6, Month 12 after surgery
Measurement of Hb1Ac | Month 3, Month 6, Month 12 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Radwan KASSIR, Dr., Principal Investigator — CHU St Etienne
Locations (1):
- Hopital Nord Chu42, Saint-Priest-en-Jarez, France